CLINICAL TRIAL: NCT04809597
Title: Study of the Activity and Role of Notch1 Signalling in Glioma
Brief Title: Does Notch Regulate Glioma Proliferation ?
Acronym: GLIONOTCH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0172
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Glioma
Keywords: pathologist-graded gliomas
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators showed in 2015 (Guichet et al) that the Notch1 pathway has an anti-proliferative role on glial brain tumors. In this project, the investigators investigated which genes downstream of Notch1 pathway activation produce the anti-proliferative effect. The investigators hypothesized that the SNAI2 and TAL1 genes act downstream of Notch1

DETAILED DESCRIPTION:
Main objectives:

To examine the expression of TAL1 and SNAI2 in protein extracts and glioma sections of different grades (glioblastomas and diffuse low-grade tumors).

To examine the effect of overexpression of Tal1 and Snai2 in high grade glioma cultures.

To show the expression of Tal1 and SNAI2 by tumor cells by FISH technique. Show that TAL1 and SNAI2 could be regulated by endothelial cells

ELIGIBILITY:
Inclusion criteria:

* Patient ≥18 years old
* Patient affected with brain glioma classified according to WHO 2016 classification

Exclusion Criteria:

* Patient who reject the study protocol
* Radiotheray or chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with brain diffuse low grade and high grade gliomas (glioblastomas)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Effect of Notch1 activation on Tal1 | 1 day
  highthroughput gene analysis (DNA arrays) with cells transduced with activated form of Notch1
Snai2 gene and protein expression | 1 day
  western blot for Tal1 and Snai2 in protein extracted from low grade and high gliomas

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Hugnot, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC